CLINICAL TRIAL: NCT00360646
Title: Idiosyncratic Liver Injury Associated With Drugs (ILIAD): A Retrospective Study
Brief Title: Drug-Induced Liver Injury (DILI) Network Retrospective
Acronym: ILIAD
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00113362; 2U01DK065176-21 (NIH); Pro00072297 (Other: Advarra); Pro00017208 (Other: original Duke IRB number)
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Drug Induced Liver Injury
Keywords: LIVER DIS; CHEM IND; Drugs; Drug induced liver injury; phenotype; cholestatic liver injury; hepatocellular liver injury; mixed liver injury; genotype
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with liver injury
- Subjects without liver injury

SUMMARY:
The purpose of this study is to establish retrospectively a nationwide registry of patients who have suffered drug-induced liver injury (DILI), and to collect, immortalize, and store serum, DNA, and lymphocytes from these patients. ILIAD will serve as a resource for subsequent mechanistic investigations into the basis of severe idiosyncratic DILI. The primary goal of the ILIAD protocol is to create: (a) a clinical database consisting of individuals who have experienced severe DILI and the relevant clinical data concerning the episode of DILI; and, (b) to create a bank of biological specimens obtained from these individuals. These biological specimens will be DNA, plasma, and immortalized lymphocytes. Immortalized lymphocytes will provide unlimited amounts of genomic DNA for study as well as living immune cells for phenotyping studies.

A secondary goal of the ILIAD protocol is to maintain a registry of cases in the ILIAD database so that they may be recontacted in the future. It is expected that this will facilitate additional studies exploring the mechanisms of DILI.

DETAILED DESCRIPTION:
Drug-induced liver injury (DILI) is the single most common reason for regulatory actions concerning drugs, including failure to gain approval for marketing, removal from the market place, and restriction of prescribing indications. DILI is also a significant cause of morbidity and mortality in many patient populations. To stimulate and facilitate research into DILI, the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) has recently established the Drug-Induced Liver Injury Network (DILIN). One of the initial projects to be conducted by the network is to retrospectively establish a nationwide registry of patients who have suffered severe idiosyncratic liver injury associated with any drugs (ILIAD) and HDS agents, and to collect, immortalize and store serum, DNA, and lymphocytes from these patients (hereafter referred to as the "ILIAD protocol"). This ILIAD protocol will serve as a resource for subsequent mechanistic investigations of the basis for susceptibility to severe idiosyncratic DILI.

The network will initially identify people who have developed DILI onset beyond 6 months of enrollment due to all drugs or HDS/CAM cases that did not meet the entrance criteria for the Prospective study.

The specific aims are as follows:

1. Establish and maintain a clinical database of these people that contains relevant clinical data.
2. Establish a bank of biological specimens (serum, DNA, and immortalized lymphocytes) prepared from cases and control in the clinical database.
3. Maintain a registry including yearly updated contact information of the subjects enrolled in the clinical database so that it is possible to recontact these individuals at a later date to offer participation in studies which are not part of the current proposal.

ELIGIBILITY:
Inclusion Criteria:

Screening Criteria

To be included in the ILIAD registry, the following criteria must be satisfied:

* The treating gastroenterologist / hepatologist or health care professional must believe that the subject suffered drug-induced liver injury;
* The subject must be alive and the date of onset of the qualifying DILI episode must have occurred on or after January 1, 1994;
* Evidence of injury that is known or suspected to be related to consumption of a drug or HDS/CAM product
* The subject is taking only one of these drugs or HDS agent(s) in the period leading up to the onset of the qualifying DILI episode;
* Have clinically important DILI defined in terms of serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (Alk Phos).
* Sufficient documentation of the event for the Causality Committee to make a determination.

Exclusion Criteria:

Subjects will be excluded according to the following criteria:

* are not willing to have medical information and blood samples taken;
* are unable to adequately give informed consent to participate in the study including the blood draw for the genetic component;
* age < 2 years old at the time of study enrollment (due to blood volume requirements).
* Have a competing cause of liver injury such as hepatic ischemia that the investigator felt to be the primary reason for the observed liver injury. Known, pre-existing autoimmune hepatitis; primary biliary cirrhosis, primary sclerosing cholangitis, or other chronic biliary tract disease. Subjects are excluded due to acetaminophen hepatoxicity or liver transplant or allogeneic bone marrow transplant prior to development of drug-CAM induced liver injury.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with liver injury ascribed to any drug or HDS/CAM agent which the DILI onset date occurred beyond six months from enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2004-09 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
maintain a registry of cases in the ILIAD database | July 2028
  maintain a registry of cases in the ILIAD database

CONTACTS AND LOCATIONS:
Overall Officials: Huiman X. Barnhart, PhD, Principal Investigator — Duke University; Robert Fontana, MD, Study Chair — University of Michigan
Locations (6):
- United States (6):
  - University of Southen California, Los Angeles, California
  - Indiana University, Indianapolis, Indiana
  - NIH Clinical Site, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Univeristy of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Thomas Jefferson, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Rochon J, Protiva P, Seeff LB, Fontana RJ, Liangpunsakul S, Watkins PB, Davern T, McHutchison JG; Drug-Induced Liver Injury Network (DILIN). Reliability of the Roussel Uclaf Causality Assessment Method for assessing causality in drug-induced liver injury. Hepatology. 2008 Oct;48(4):1175-83. doi: 10.1002/hep.22442. PMID 18798340
- See also: Multi-center, Longitudinal Study of Drug-and-CAM-Induced Liver Injury — https://dilin.org/
- See also: The National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) is part of the National Institutes of Health (NIH) — http://www.niddk.nih.gov